CLINICAL TRIAL: NCT01048762
Title: Multidisciplinary Rehabilitation After Cancer Pulmonis Operation - a Randomized Controlled Trial
Brief Title: Multidisciplinary Rehabilitation After Cancer Pulmonis Operation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); The Danish Cancer Foundation - Research Department - North Region (Unknown); University of Aarhus (Other)
Responsible Party: Principal Investigator, Barbara C. Brocki, Physiotherapist, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tp.afd-001
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Pulmonary Cancer
Keywords: pulmonary cancer; radically operated; exercise training; dyspnea counseling; quality of life; physical therapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Exercise; Resistance Training; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- supervised exercise training (Active Comparator): Intervention: supervised exercise training and dyspnea counseling in groups for 10 weeks Instruction on home based exercise training
  Interventions: Other: physical exercise and dyspnoea counseling; Other: home training
- one instruction on homebased exercises (Sham Comparator): One instruction on home based exercise training and dyspnea management
  Interventions: Other: home training

INTERVENTIONS:
Other: physical exercise and dyspnoea counseling — Exercise training in group, 1 hour once a week for 10 weeks, based om aerobic exercises 60-80% of VO2 max (Borg 11-12), resistance training and dyspnea counseling. Participants are urge to exercise training for at least twice a week.
  Other Names: aerobic exercise training and resistance training; dyspnea counseling; training in groups
  Arms: supervised exercise training
Other: home training — one instruction in home based exercise training
  Other Names: home based exercises

SUMMARY:
The purpose of this investigation is to determine the effects of exercise training on quality of life and physical capacity, 3 months and 1 year after radical operation for pulmonary cancer.

DETAILED DESCRIPTION:
Patients who are radically operated for pulmonary cancer report suffering from respiratory problems, mostly dyspnoea, 5 years after operation. Dyspnoea restricts their physical capability and leads to poorer physical, social and mental wellbeing. The effects of training programs on physical and mental wellbeing for cancer patients are well documented. Most of the studies are though performed on patients suffering from breast, colon and prostate cancer. There are only few studies addressing patients with pulmonary cancer. They are mostly focused on short term effects of exercise training on quality of life, with no control group included in the trials. These studies target patients after different forms for treatment, including surgery, chemotherapy and radiation. There is no data referring to quality of life of patients who are radically operated for pulmonary cancer.

Comparison: multidisciplinary group intervention consisting of exercise training and dyspnoea counseling, 10 times, once a week, compared with one instruction in exercise training and dyspnoea counseling. Exercise training is given by a physiotherapist. Both groups receive in addition standard treatment, which is up to 3 counseling sessions with a nurse.

ELIGIBILITY:
Inclusion Criteria:

* patients who are radically operated for pulmonary cancer at Aalbor Hospital, Aarhus University Hospital

Exclusion Criteria:

* not radically operated
* cannot speak and read Danish
* cannot cooperate in tests due to poor mental health
* patients who undergo rehabilitation at other centres
* cannot perform walking test due to physical impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-02; Primary Completion 2010-01 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Changes in selv reported quality of life and physical capacity 4 months after inclusion measured by SF-36 and 6MWT | 4 months after inclusion

SECONDARY OUTCOMES:
Changes in selv reported quality of life and physical capacity 1 year after inclusion, measured by SF-36 and 6MWT | 1 year after inclusion
Changes in lungfunction 4 months and 1 year after inclusion (FEV1, FVC and FEV1/FVC) | 4 months and 1 year after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Vitautas Nekrasas, Chief doctor, Study Chair — Department of Cardiothoracic Surgery, Centre for Cardiovascular Research, Aalborg Hospital, Aarhus University Hospital
Locations (1):
- Department of Rehabilitation, Aalborg Hospital, Aarhus University Hospital, Aalborg, Denmark